CLINICAL TRIAL: NCT03507491
Title: AflacST1603: a Phase 1 Study Using Nab-paclitaxel (Abraxane®) in Combination with Gemcitabine for Pediatric Relapsed and Refractory Solid Tumors
Brief Title: Nab-paclitaxel in Combination with Gemcitabine for Pediatric Relapsed and Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, William T Cash, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00098777
Record Dates: First submitted 2018-03-22; First posted 2018-04-25 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Cancer
Keywords: Pediatric; Sarcoma; Neuroblastoma; Ewing sarcoma; Osteosarcoma; Rhabdomyosarcoma; Wilms tumor; Hepatoblastoma; Adolescent and young adult; Germ cell tumor
MeSH Terms: conditions — Neoplasms; Sarcoma; Neuroblastoma; Sarcoma, Ewing; Osteosarcoma; Rhabdomyosarcoma; Wilms Tumor; Hepatoblastoma; Neoplasms, Germ Cell and Embryonal | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gemcitabine + Nab-paclitaxel (Experimental): Participants receiving gemcitabine and nab-paclitaxel for refractory and/or relapsed solid tumors of childhood.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine will be administered intravenously once weekly over 60 minutes every 3 out of four weeks. The dose of gemcitabine will start at 675 mg/m2/dose. If the MTD has been exceeded at the Dose Level 1, then the subsequent cohort of participants will be treated with gemcitabine at a dose of 500 mg/m2/dose (Dose Level 0).
  Other Names: Gemzar
Drug: Nab-paclitaxel — Nab-Paclitaxel will be administered intravenously over 30 minutes once weekly every 3 out of 4 weeks. Nab-paclitaxel will be administered prior to administration of gemcitabine. The starting dose of nab-paclitaxel will be 180 mg/m2/dose (dose level 1). Dose levels for subsequent groups of subjects are 210 mg/m2/dose (for dose level 2) and 240 mg/m2/dose (for dose level 3).
  Other Names: Abraxane

SUMMARY:
This is a research study for people who have a solid tumor that was not effectively treated by conventional therapy or for which there is no known effective therapy. This is a phase I study of a drug called nab-paclitaxel used together with gemcitabine. Gemcitabine and nab-paclitaxel will be given intravenously, once a week for 3 out of 4 weeks, for a 28-day cycle.

The goals of this study are:

* To find the highest dose of nab-paclitaxel that can be safely given in combination with gemcitabine without causing severe side effects
* To learn what kind of side effects nab-paclitaxel given in combination with gemcitabine can cause
* To learn more about the pharmacology (how the body handles the drug) of nab-paclitaxel given in combination with gemcitabine
* To evaluate tumor tissue for levels of certain proteins that may help with predicting who will benefit most from treatment with nab-paclitaxel
* To determine whether nab-paclitaxel given in combination with gemcitabine is a beneficial treatment for relapsed and/or refractory solid tumors

DETAILED DESCRIPTION:
Relapsed and refractory non-central nervous system (non-CNS) solid tumors have poor outcomes, and novel therapies are needed. Many relapsed/refractory solid tumor patients desire further therapy; however, they often wish to also preserve a high quality of life. Thus therapeutic strategies that offer relatively minimal treatment-related toxicities are also desirable. The combination of gemcitabine, a pyrimidine analog, and docetaxel, an antimitotic taxane, is an attractive combination because of non-overlapping toxicities. This combination has shown activity and tolerability in adult Phase II trials for solid tumors. Favorable experiences with this regimen in pediatrics have been described retrospectively by several institutions. Nab-paclitaxel is an albumin-bound, solvent-free taxane that allows higher dosing and shorter infusion duration than solvent-bound taxanes (docetaxel and paclitaxel) by removing exposure to toxic solvent carriers. Albumin binding of the agent also increases drug delivery to tumors through increased albumin-initiated transcytosis, and may also increase tumoral accumulation of drug through binding of secreted protein acidic and rich in cysteine (SPARC). The combination of gemcitabine and nab-paclitaxel has been studied extensively in adults with pancreatic adenocarcinoma, with the combination providing superior outcomes to treatment with gemcitabine alone. There is also preclinical evidence of potent anti-tumor activity of nab-paclitaxel alone and in combination with gemcitabine in pediatric solid tumor models. Therefore, the researchers hypothesize that the combination of nab-paclitaxel with gemcitabine will improve the anti-tumor efficacy observed with gemcitabine/docetaxel in relapsed/refractory solid tumors.

This is a Phase 1 study of nab-paclitaxel in combination with gemcitabine for children, adolescents, and young adults with relapsed or refractory non-central nervous system (CNS) solid tumors in which the researchers will define toxicity, pharmacokinetics, and evaluate SPARC expression in pediatric tumors as a biomarker of disease response.

Nab-paclitaxel will be administered intravenously (IV) once weekly on days 1,8, and 15 of a 28 day cycle. The starting dose of nab-paclitaxel will be 180 mg/m2/dose which is 75% of the pediatric, single agent MTD of 240 mg/m2/dose. The researchers will then dose escalate up to 240 mg/m2/dose. Dose Level 1 of the protocol prior to Amendment 2 utilized nab-paclitaxel at 180 mg/m2/dose and gemcitabine and 1000 mg/m2/dose given on days 1, 8, and 15 of 28 day cycles. The study enrolled 5 patients at Dose Level 1 and two patients experienced hematologic dose limiting toxicities (DLTs). Amendment 2 decreases the starting dose of gemcitabine on Dose Level 1 to 675 mg/m2/dose on days 1, 8, and 15 of the 28 day cycle. If Dose Level 1 is tolerated, then the dose of nab-paclitaxel will escalated on subsequent dose levels. If two or more participants experience DLTs at Dose Level 1, then the study will de-escalate to Dose Level 0 by decreasing the gemcitabine dose to 500 mg/m2/dose IV days 1, 8, and 15. If Dose Level 0 is tolerated, then a dose escalation of nab-paclitaxel will occur.

Participants may continue on therapy until there is evidence of progressive disease or toxicity that requires removal from therapy. Therapy may otherwise continue for up to 24 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥ than 6 months and ≤ 30 years of age at the time of study enrollment.
* Subjects must have had histologic verification of a malignancy at original diagnosis or relapse.

  * All subjects with relapsed or refractory solid tumors are eligible, excluding primary CNS tumors.
  * Patients with solid tumors and a history of intraparenchymal CNS disease are eligible if their CNS disease was treated surgically or with radiotherapy and stable with no recurrent lesions for at least 3 months from the start of protocol therapy.
  * Newly diagnosed patients with ≤15% chance of cure if given standard-of-care chemotherapy are eligible. (Prognosis to be determined at the discretion of the treating physician.)
* Subjects must have either measurable or evaluable disease.
* Karnofsky ≥ 60 for subjects > 16 years of age and Lansky ≥ 50 for subjects ≤ 16 years of age. Subjects who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Subjects must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy.

  * At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea).
  * At least 14 days after the last dose of a long-acting growth factor (e.g. Pegfilgrastim) or 7 days for short acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
  * At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
  * ≥ 42 days must have elapsed from last dose of any type of cellular therapy (e.g. modified T cells, natural killer (NK) cells, dendritic cells, etc.)
  * ≥ 21 days must have elapsed from the last dose of interleukins, interferon or cytokines (other than Hematopoietic Growth Factors).
  * ≥ 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to Grade ≤ 1.
  * At least 14 days after local palliative radiation therapy (XRT) (small port); 6 weeks must have elapsed since treatment with therapeutic doses of iodine-131 metaiodobenzylguanidine (131I-MIBG); At least 42 days must have elapsed if other substantial bone marrow (BM) radiation.
  * No evidence of active graft vs. host disease and at least 84 days must have elapsed after transplant and 42 days for autologous stem cell infusion after 131I-MIBG therapy.
  * Patients who have previously received a taxane, including nab-paclitaxel, or a nucleoside analogue, including gemcitabine, are eligible as long as they have not received gemcitabine in combination with nab-paclitaxel.
  * ≥72 hours must have elapsed since the last administration of medical cannabis and cannabidiol (CBD Oil).
  * ≥30 days must have elapsed since the last dose of any agents not specified above. For agents with an uncertain washout period or for any questions or uncertainty the study PI should be notified.
* Adequate bone marrow function defined as:

  * For subjects with solid tumors without known bone marrow involvement: Peripheral absolute neutrophil count (ANC) ≥ 750/mm3. Platelet count ≥ 75,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
  * Subjects with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts of peripheral absolute neutrophil count (ANC) ≥ 750/mm3 and platelet count ≥ 75,000/mm3 (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions). These subjects will not be evaluable for hematologic toxicity. At least 5 of every cohort of 6 patients must be evaluable for hematologic toxicity for the dose-escalation part of the study. If dose-limiting hematologic toxicity is observed, all subsequent subjects enrolled must be evaluable for hematologic toxicity.
* Adequate renal function defined as:

  * Creatinine clearance or radioisotope glomerular filtration rate (GFR) 70ml/min/1.73 m^2 or
  * A serum creatinine based on age/gender using threshold creatinine values derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the Centers for Disease Control and Prevention (CDC).
* Adequate liver function defined as:

  * Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age
  * Serum glutamic pyruvic transaminase (SGPT) (ALT) ≤ 5 x the ULN. For the purpose of this study, the ULN for SGPT is 45 U/L.

Exclusion Criteria:

* Female patients who are pregnant are ineligible for study. Lactating females are not eligible unless they have agreed not to breastfeed their infants from the time of informed consent through the duration and at least 1 month following the last dose of investigational agent. Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained. Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method from the time of informed consent through the duration and for 1 month following the last dose of investigational agent. The definition of an effective contraceptive method will be at the discretion of the institutional investigator.
* Patients taking any the following concomitant medications are not eligible:

  * Subjects who are currently receiving another investigational drug.
  * Subjects who are currently receiving other anti-cancer agents.
  * Subjects who are receiving cyclosporine, tacrolimus, or other agents to prevent graft-versus-host disease post bone marrow transplant.
  * Subjects using medications which interfere with CYP3A4 and CYP2C8 metabolism, which metabolize nab-paclitaxel. Paclitaxel is metabolized by CYP3A4 and CYP2C8, so strong inhibitors or inducers of these enzymes should be avoided.
* Patients with any of the following adverse events at the time of enrollment are not eligible:

  * Grade ≥ 2 Motor, sensory or peripheral neuropathy. This does not apply to patients with neuropathic symptoms related to tumor or prior therapy, i.e. surgery or radiation. Patients with mild neuropathy well controlled with medications are eligible.
  * Grade ≥3 Hyponatremia (serum Na ≤ 130 mmol/L)
* Subjects who have an uncontrolled infection are not eligible.
* Subjects who have received prior solid organ transplantation are not eligible.
* Subjects who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Maximum dose tolerated of nab-paclitaxel | Up to Day 28
  The maximum tolerated dose (MTD) of nab-paclitaxel administered intravenously weekly every 3 of 4 weeks in combination with gemcitabine in children with refractory/relapsed non-CNS solid tumors will be determined. The MTD is empirically defined as the highest dose level at which there is no more than one patient experiencing a dose-limiting toxicity (DLT) and the next higher dose level has been determined to be too toxic. The MTD will be determined during Cycle 1 (each cycle is 28 days)
Toxicity of nab-paclitaxel | Up to 96 weeks
  The toxicities of nab-paclitaxel in combination with gemcitabine administered intravenously weekly every 3 of 4 weeks will be determined. All toxicities observed will be summarized in terms of type (organ affected or laboratory determination), severity (by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0), and attribution. Data on toxicities will be collected during the entire time a participant is in the study (up to 24 cycles, each cycle is 28 days).

SECONDARY OUTCOMES:
Antitumor activity of nab-paclitaxel | Up to 96 weeks
  The antitumor activity (tumor growth) of nab-paclitaxel in combination with gemcitabine will be preliminarily defined, within the confines of a Phase 1 study.
Change in secreted protein acidic and rich in cysteine (SPARC) expression | Up to 96 weeks
  The expression of SPARC in tumor tissue from pediatric solid tumors will be evaluated. Archived tumor samples obtained as part of routine subject care will be evaluated for immunohistochemical expression of SPARC. Samples will be evaluated from all surgical procedures to evaluate if expression of these factors changes over time and can predict tumor responsiveness to therapy. Specifically, samples from diagnosis, post-therapy resection, and relapse (when performed for clinical reasons) will be evaluated.
Blood concentrations of paclitaxel | Up to Day 3
  Blood samples will be collected for the first dose (Cycle 1, Day 1) from all patients on study to analyze paclitaxel concentrations in blood. Blood samples will be obtained on Day 1 of Cycle 1 at 1-2 min prior to end of infusion, and 0.25, 1, 3, 5, 7, 24, and 48 hours after end of the nab-paclitaxel infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cash, MD, MSc, Study Chair — Emory University; Jonathan Metts, MD, Study Chair — Johns Hopkins All Children's Hospital
Locations (4):
- United States (4):
  - Children's Hospital Colorado, Aurora, Colorado
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Chilldren's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Mercy Hospital, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No